CLINICAL TRIAL: NCT04785534
Title: Patient-Centered Liver Cancer Prevention in the Houston Community Screening for Predictors of Fibrosis and Cirrhosis
Brief Title: Surveys, Blood Testing, and Fibroscan in Screening for Liver Fibrosis and Liver Cirrhosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2019-0978; NCI-2021-00214 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-02-04; First posted 2021-03-08 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Liver and Intrahepatic Bile Duct Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (survey, biomarker analysis, fibroscan) (Experimental): Patients complete surveys over 10-15 minutes, and undergo blood testing, clinical evaluation, and fibroscan at baseline.
  Interventions: Other: Clinical Evaluation; Other: Laboratory Biomarker Analysis; Procedure: Liver Ultrasonographic Elastography; Other: Survey Administration

INTERVENTIONS:
Other: Clinical Evaluation — Undergo clinical evaluation
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Liver Ultrasonographic Elastography — Undergo fibroscan
  Other Names: Fibroscan; TE; Transient Elastography; VCTE; Vibration-Controlled Transient Elastrography
Other: Survey Administration — Complete survey

SUMMARY:
This clinical trial studies the use of surveys, blood testing, and fibroscan in screening for liver fibrosis and liver cirrhosis in new or existing patients of the HOPE clinic seeking usual clinical care. Fibroscan is an imaging procedure of the liver which uses a probe like an ultrasound. Information gathered from this study may help researchers learn more about how to prevent or find liver cancer in patients who are currently receiving care at the HOPE clinic. Early detection of liver cancer may improve survival.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the sensitivity of the modified Center for Disease Control (CDC) hepatitis survey in diagnosing chronic hepatitis B virus (HBV) among HOPE clinic patient.

SECONDARY OBJECTIVES:

I. To estimate the sensitivity of the modified CDC hepatitis survey in identifying chronic active hepatitis C virus (HCV) infection among HOPE clinic patients.

II. To estimate the sensitivity of fibrosis serum biomarkers, non-alcoholic fatty liver disease fibrosis score (NFS), fibrosis-4 index (FIB-4), and fatty liver index (FLI) in detecting fibrosis (fibroscan result >= F2) among HOPE clinic patients with metabolic conditions.

III. To estimate the sensitivity of the Alcohol Use Disorder Identification Test Alcohol Consumption (AUDIT-C) in identifying fibrosis (fibroscan result >= F2) among HOPE clinic patients.

IV. To estimate the sensitivity of the AUDIT-10 survey in identifying fibrosis (Fibroscan result >= F2) among Hope Clinic patients who scored >= 4 for men or >= 3 for women on the AUDIT-C.

V. To estimate the specificity and accuracy of each of these risk factor screening tools in HOPE clinic patients.

VI. To estimate the prevalence of fibrosis and cirrhosis risk factors among HOPE clinic patients.

EXPLORATORY OBJECTIVES:

I. To explore factors associated with each fibrosis/cirrhosis risk factor. II. To investigate differential diagnostic accuracy of screening methods by fibrosis severity.

III. To evaluate the diagnostic performance of each dichotomized biomarker (NFS, FIB-4, and FLI) separately and assess biomarker optimal cutpoints for identifying fibrosis in the study population.

OUTLINE:

Patients complete surveys over 10-15 minutes, and undergo blood testing, clinical evaluation, and fibroscan at baseline.

After completion of study, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old
* Must be a new or existing patient of the HOPE clinic seeking usual clinical care
* Must be able to speak and read English or a language other than English for which there is a translator available on site at the HOPE clinic

Exclusion Criteria:

* Known pregnancy at time of recruitment. The HOPE clinic will ask the female patients if they are pregnant, will ask the participants for their last menstrual period (LMP), and/or they will use the urine pregnancy test (UPT) results in their electronic medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Positive hepatitis B surface antigen test result | At baseline
  The presence of at least one risk factor for hepatitis B virus (HBV) on the screening questionnaire will indicate a positive (versus negative) screening for HBV infection.

SECONDARY OUTCOMES:
Positive anti-hepatitis C virus (HCV) test result | At baseline
  Will assess positive anti-HCV test result AND either 1) detectable HCV ribonucleic acid, or 2) history of HCV infection and past anti-HCV treatment. Will estimate the prevalence and exact binomial 95% confidence intervals for each of the fibrosis and cirrhosis risk factors examined in this study. For each risk factor, we will first present a cross tabulation of the dichotomous screening test result by the dichotomous gold standard result. To evaluate the performance of each screening method, will calculate point estimates and 95% confidence intervals for the sensitivity, specificity, likelihood ratio, and diagnostic odds ratio.
Fibroscan result >= F2 | Up to 3 months
  Will estimate the prevalence and exact binomial 95% confidence intervals for each of the fibrosis and cirrhosis risk factors examined in this study. For each risk factor, we will first present a cross tabulation of the dichotomous screening test result by the dichotomous gold standard result. To evaluate the performance of each screening method, will calculate point estimates and 95% confidence intervals for the sensitivity, specificity, likelihood ratio, and diagnostic odds ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica P Hwang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT04785534/ICF_000.pdf